CLINICAL TRIAL: NCT06762054
Title: Investigating the Optimal Management of Dolutegravir Resistance: a Multi-country Cohort Study
Brief Title: Investigating the Optimal Management of Dolutegravir Resistance
Status: Recruiting | Type: Observational
Sponsor: University of Nairobi (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); Muhimbili University of Health and Allied Sciences (Other); SolidarMed (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Loice Achieng Ombajo, Chief Investigator, University of Nairobi
Other Study IDs: Ndovu Cohort Study
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: HIV-1-infection
Keywords: HIV; Dolutegravir; Treatment failure; Drug resistant mutations; Dolutegravir resistance; Re-suppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples stored at baseline and at all timepoints where a viral load test is conducted for possible HIV drug resistance testing (DRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Continue DTG-based antiretroviral therapy — Participants will continue on DTG-based ART after enrollment for up to 12 months
Behavioral: Enhanced adherence counselling — Participants with VL ≥200 copies/mL will undergo enhanced adherence counselling

SUMMARY:
The goal of this study is to address the gap in published data on viral suppression among people meeting the criteria for virologic failure on dolutegravir (DTG)-based ART regimens without a change in regimen. The study will also assess the emergence of DTG-associated drug-resistant mutations and their impact on viral suppression.

DETAILED DESCRIPTION:
BACKGROUND:

The majority of people living with HIV (PLWH) on first line antiretroviral therapy (ART) in low and middle-income countries are on dolutegravir (DTG)-containing regimens. Different countries have adopted different approaches in the management of people on DTG-based first line ART with repeat HIV viral load (VL) of > 1,000 copies/mL after 3 months of enhanced adherence counseling. For example, Kenya recommends a drug resistance test (DRT) to guide on switch and the optimal second line regimen; Mozambique and Tanzania recommend switch to 2 nucleoside reverse transcriptase inhibitors (NRTIs) and protease inhibitors (PIs) without drug resistance testing; South Africa does not recommend switch from DTG or DRT for those who are on first-line DTG-containing regimens within the first 2 years of treatment, after which management is guided by possible DRT and expert opinion. The World Health Organization has recognised the role of drug resistance testing (DRT) in a treatment failure algorithm for people living with HIV receiving DTG-based treatment to minimise unnecessary switches from this regimen. The switch to PI has disadvantages including higher cost, higher pill burden, less convenient administration (often should be taken with food), more potential drug-drug interactions, poorer tolerability and more long-term toxicities.

OBJECTIVE:

To assess viral suppression rate following enhanced adherence counseling among people on DTG-based ART who have sustained viraemia (≥ 1,000 copies/mL) after at least six months on ART.

METHODS:

This is a multi-country observational prospective cohort study over 12 months describing HIV-1 viral suppression in people with high viral load (≥ 1,000 copies/mL) after at least six months on DTG-based ART. The Study targets to enrol 6,600 participants in Kenya, Mozambique, Tanzania and Lesotho. Study visits and VL testing will take place at enrolment and then every 3 months for up to 12 months during the active follow-up period for participants who do not achieve viral suppression < 200 copies/mL. During each visit, protocol-specified enhanced adherence counseling and assessment/management of other causes of viremia will continue for at least 3 sessions. For participants who achieve the primary outcome of HIV-1 RNA < 200 copies/mL during the active follow-up period, a repeat VL will be performed after 3 months; outcomes from routinely collected program data (viral load, loss to follow-up, death) will be collected 12-24 months from enrolment to assess durability of suppression among this group. The investigators will estimate the viral suppression at 6 and 12 months using a generalized linear regression model with binomial distribution as well as assess for predictors of achieving suppression, development of DTG-associated drug resistance mutations (DRMs), and development of opportunistic infections using logistic regression models. Participants will also be assessed for eligibility to enrol into a nested randomized clinical trial (RCT) on management of people who develop DRMs during the cohort study (Ndovu RCT; see separate protocol).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent (assent as appropriate and legal guardian consent if < 18 years)
* Age ≥ 1 years
* Documented HIV-1 infection as confirmed by national HIV testing standards at the respective study sites
* On a DTG-based ART regimen for at least six months
* Most recent HIV-1 RNA ≥ 1,000 copies/mL within 3 months prior to enrolment, taken after at least 6 months on current ART regimen

Exclusion Criteria:

* Has switched ART regimen for confirmed or suspected HIV treatment failure while on a PI- or INSTI-based regimen
* Any reason which, in the investigator's opinion, will significantly prevent the collection of viral load levels such as relocation to another area outside of the trial sites or imminent death
* Concomitant NNRTI or PI while on DTG

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited without advertisement from the pool of patients receiving routine outpatient HIV care at the study sites and at surrounding HIV clinics in 8 central study sites in Kenya, 1 central study site in Tanzania (enrolling from surrounding care and treatment centres in Dar es Salaam), 6 study sites in Mozambique, and 5 study sites in Lesotho. The target sample size for this study is 6,600 participants. Participants who develop DTG-associated DRMs during cohort follow-up will be assessed for eligibility into a clinical trial assessing the optimal management of people who develop drug resistance to DTG-based ART (Ndovu RCT).
Sampling Method: Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Viral suppression rate | 12 months
  Viral suppression rate following enhanced adherence counseling

SECONDARY OUTCOMES:
Time to viral suppression | 12 months
  Time to HIV-1 viral suppression to < 200 copies/mL
Viral suppression by age strata | 12 months
  Viral load suppression rate by age strata: 1-9, 10-19, ≥20, 20-24, 25-34, 35-44, and ≥45 years old
Viral suppression by viral load strata | 12 months
  Viral load suppression by viral load strata: 1,000-99,999, and ≥100,000 copies/mL
Viral suppression by sex at birth | 12 months
  Viral load suppression based on participant's sex
Viral suppression by nucleoside/nucleotide reverse transcriptase inhibitor (NRTI) | 12 months
  Viral load suppression based on the NRTI component of the antiretroviral regimen
Durability of suppression | 12 to 24 months
  Durability of suppression at 3 months from first viral load of <200 copies/mL
Incidence of drug resistant mutations (DRMs) | 12 months
  Incidence of treatment-emergent drug resistant mutations
Drug resistant mutations patterns | 12 months
  Drug resistant mutations (DRM) patterns (dolutegravir (DTG)-associated DRMs with or without concomitant nucleoside reverse transcriptase inhibitors drug resistant mutations) associated with sustained non-suppression or viral rebound after suppression
Predictors of development of dolutegravir (DTG)-associated drug resistant mutations | 12 months
  What are the predictors of development of dolutegravir (DTG)-associated drug resistant mutations
Time from viraemia to drug resistant mutations | 12 months
  Time from first detected viraemia to development of dolutegravir (DTG)-associated drug resistant mutations

CONTACTS AND LOCATIONS:
Overall Officials: Loice A Ombajo, MMed, MSc, Principal Investigator — University of Nairobi
Locations (9):
- Kenya (3):
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
  - Bomu Hospital, Mombasa
  - Kenyatta National Hospital, Nairobi
- Lesotho (2):
  - Butha-Buthe District Hospital, Butha-Buthe
  - Mokhotlong District Hospital, Mokhotlong
- Mozambique (3):
  - CS Ponta Gea, Beira, Sofala
  - CS Machava II, Maputo
  - CS Ndlavela, Maputo
- MUHAS Clinical Trial Unit, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the individual patient data (IPD) that underlie the results reported after de-identification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after publication of the final manuscript and for a period of 36 months
Access Criteria: Access to IPD will be subject to the University of Nairobi data sharing requirements. Written requests should be submitted to the Principal Investigator providing a brief description of the individual or group making the request and detailing the reason for the same. Prior to sharing the data, the requestor will be required to sign a data access and sharing agreement.